CLINICAL TRIAL: NCT02726828
Title: Effects of Intrathecally Administered Ketamine, Morphine and Their Combination in Patients Undergoing Major Abdominal Cancer Surgery
Brief Title: intrathecaم Ketamine, Morphine and Both for Lower Abdominal Cancer Surgery Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Lecturer of anesthesia, icu, and pain management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 165
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group I: morphine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.3 mg morphine in 1 ml volume intrathecally.
  Interventions: Drug: intrathecal morphine
- group II: ketamine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.1 mg/kg ketamine in 1ml volume intrathecally.
  Interventions: Drug: intrathecal ketamine
- group III: morphine + ketamine group (Active Comparator): patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.3 mg morphine plus 0.1 mg/kg of Ketamine in 1 ml volume intrathecally.
  Interventions: Drug: intrathecal morphine + ketamine

INTERVENTIONS:
Drug: intrathecal morphine — patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.3 mg intrathecal morphine1 ml volume.
  Arms: group I: morphine group
Drug: intrathecal ketamine — patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.1 mg/kg intrathecal ketamine in 1ml volume.
  Arms: group II: ketamine group
Drug: intrathecal morphine + ketamine — patients received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and intrathecal morphine + ketamine 0.3 mg and 0.1 mg/kg respectively in 1 ml volume.
  Arms: group III: morphine + ketamine group

SUMMARY:
this study investigates the analgesic efficacy and other possible effects of ketamine, morphine, and both together when administered intrathecally for control of postoperative pain following lower abdominal cancer surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) I-III patients.
* aged 30-50 years.
* scheduled for major abdominal cancer surgery.

Exclusion Criteria:

* Patients with a known allergy to the study drugs.
* significant cardiac, respiratory, renal or hepatic disease.
* coagulation disorders.
* infection at or near the site of intrathecal injection.
* drug or alcohol abuse.
* BMI > 30 kg/m2.
* psychiatric illnesses that may interfere with perception and assessment of pain.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) scores | 24 hours postoperative
  postoperative pain measured by this score.
time to first analgesic request | 24 hours postoperative
  the time passed till the first request of rescue analgesia by the patients
total analgesic consumption | 24 hours postoperative
  the total amount of rescue analgesic drug used allover follow up period

SECONDARY OUTCOMES:
side effects | 24 hours postoperative
  the type and rate of incidence of side effects during the follow up period

IPD SHARING:
Plan to Share IPD: Undecided